CLINICAL TRIAL: NCT03027986
Title: Evaluation of a Postural Rehabilitation Program Based on Sensory-motor Control in Men With Urinary Incontinence After Prostatectomy
Acronym: PROTOMEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/210/HP
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Urinary Incontinence; Prostate Cancer
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postural rehabilitation program based on sensory-motor control (Experimental)
  Interventions: Behavioral: postural rehabilitation program
- Standard physiotherapy (No Intervention)

INTERVENTIONS:
Behavioral: postural rehabilitation program — This program is based on sensory-motor control
  Arms: postural rehabilitation program based on sensory-motor control

SUMMARY:
Urinary incontinence (UI) is defined by the International Continence Society as "any involuntary loss of urine complained by the patient". The anatomical and histological specificities of the pelvic floor muscles (PFM) give them a key role in the control of urination but also in the control of postural stability. These activities are involuntary automatisms and the mechanisms that lead to post-prostatectomy stress urinary incontinence are not only due to the loss of voluntary contraction of the pelvic floor muscles. The mechanisms that lead to UI are more complex and may involve the loss of efficacy of all deep muscle stabilizing lumbo-pelvic region. Rehabilitation of pelvic floor muscles is recommended in the treatment of urinary incontinence after prostatectomy (Grade A), but there is a lack of evidence to define the best treatment regimen for PFM rehabilitation.

Two kinds of PFM rehabilitation are are commonly practiced by specialized physiotherapists.

* The first one is made in individual box, in supine position. By analytic contractions of the PFM, (exercises of Kegel type) +/- associated with an instrumental biofeedback. This method used voluntary contractions of MPP.
* The second is realized in various positions following a gravity progression, in individual and /or common room. This technique aims to restore a stabilization of the entire lumbo-pelvic region by postural recruitment involving synergistic contractions of the PFM.

These trials propose to compare these two rehabilitation programs on populations with postoperative follow-up of more than 12 months.

We chose to objectify the urine leaks with the pad test (weighing of the protections urinary over a period of 3 times 24h) which will be our main evaluation criterion. The home test pad of 3 times in 24 hours has been used by numerous studies and its reproducibility and reliability are established.

Urinary incontinence is a recognized factor of sedentary lifestyle, fatigue, impaired mental health and decreased of physical fitness. We therefore wish to observe these parameters for each of our two randomized groups

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male
* Between the age of 18 and 78 years
* Patient who underwent prostatectomy more than 12 months ago but less than 10 years
* 3x24h pad test over or equivalent to 10 grs
* Persistent urinary incontinence beyond 12 month following prostatectomy
* Patient affiliated to social security
* Patient who submitted non-opposition for participation in the study

Exclusion Criteria:

* Patients who underwent prostatectomy or other visceral surgery less than one year ago
* Patient who underwent surgical treatment of urinary incontinence
* Patient with urinary incontinence less than 10g
* Surgery considered within two years of inclusion
* Radio, hormone, or chemotherapy cured or in progress
* Anticholinergic treatment less than 3 months ago
* Patient with neurological or bladder disorders potentially involved in incontinence disorders
* Vestibular or psychiatric pathology making limitations to carry out all the examinations provided for in the protocol
* Patient unable to complete the planned 15 visits to physiotherapist
* Patient participating in another clinical trial

Ages: 18 Years to 78 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — this medical condition for participation is patient with a prostatectomy
Enrollment: 116 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Difference from baseline in urine leakage | 6 months
  urine leakage will be measured using pad test

SECONDARY OUTCOMES:
Difference from baseline in The Berg balance scale test | 6 months
  The Berg balance scale test evaluating the quality of static and dynamic motor control.
Difference from baseline in quality of life | 6 months
  quality of life is based on EORTC QLQ C30

CONTACTS AND LOCATIONS:
Overall Officials: Benoît STEENSTRUP, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No